CLINICAL TRIAL: NCT04572386
Title: Clinical Performance of Low Technique Sensitive Self-cured Universal Adhesive Versus Light Cured Universal Adhesive in Patients With Non-carious Cervical Lesions (NCCLs): 18 Month Randomized Clinical Trial
Brief Title: Clinical Performance of Low Technique Sensitive Self Cured Universal Adhesive Vrs Light Cured Universal Adhesive in Patients With (NCCLs): 18 m RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aya Gamal ashour (Other)
Responsible Party: Sponsor-Investigator, Aya Gamal ashour, principle investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: gsda.1986.2
Record Dates: First submitted 2020-09-11; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Non Carious Cervical Lesion
Keywords: universal bond; NCCls; 3m single bond universal; Palfique, Tokuyama, Japan; self cure; non carious cervical lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Light cure universal bond (Active Comparator): light cured 3m single bond universal
  Interventions: Other: light cure 3m single bond universal bond
- self cure universal bond (Active Comparator): self-cure universal bond (Palfique, Tokuyama, Japan)
  Interventions: Other: Self-cure universal bond (Palfique, Tokuyama, Japan)

INTERVENTIONS:
Other: light cure 3m single bond universal bond — light -cure universal bond
  Arms: Light cure universal bond
Other: Self-cure universal bond (Palfique, Tokuyama, Japan) — Self-cure universal bond with no light cure
  Arms: self cure universal bond

SUMMARY:
This study will be conducted to evaluate the clinical performance of self-cured adhesive versus light cured universal adhesive in non-carious cervical lesions (NCCL) resin composite restorations after 18 month

ELIGIBILITY:
Inclusion Criteria:

* particepant with age rang 18-55
* particepant with non carious cervical lesion

Exclusion Criteria:

* particepant outside age rang
* particepant with periodontal problem that might affect the teeth to be treated

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Number of fracture restoration | 18 month
  Frist visual evaluation to ensure that there is no complete loss of retention of the restoration then tactile evaluation will be done using probe tip that will be held gently at right angle to the labial surface and move from restoration to tooth and vice versa to insure no rocking /fracture /ditching in the restoration following FDI criteria ( first visually for total loss .followed by tactile inspection using fdi prob for any fracture /rocking or loss of retention
number of restoration with retention loss | 18-month
  Frist visual evaluation to ensure that there is no complete loss of retention of the restoration then tactile evaluation will be done using probe tip that will be held gently at right angle to the labial surface and move from restoration to tooth and vice versa to insure no rocking /fracture /ditching in the restoration following FDI criteria

SECONDARY OUTCOMES:
Number of restoration with change in colour or texture | 18 month
  Evaluation will be done visually following FDI criteria to ensure no change in colour or texture of the restoration
Number of restoration caused biological harm | 18 month
  Evaluation will be done following FDI criteria using FDI prob to ensure no change in restoration that caused any harm to the health of biological strucure

IPD SHARING:
Plan to Share IPD: Undecided